CLINICAL TRIAL: NCT01806103
Title: Reducing Inappropriate Prescribing of Antibiotics by Primary Care Clinicians
Brief Title: Antimicrobial Stewardship for Primary Care Pediatricians
Acronym: PARTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-007305; HHSA2900200710013 (Other Grant/Funding Number: AHRQ HHSA2900200710013)
Record Dates: First submitted 2013-02-04; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Acute Sinusitis; Streptococcal Pharyngitis; Pneumonia; Viral Infection
Keywords: antimicrobial stewardship program; inappropriate prescribing of antibiotics; physician prescribing; antibiotic prescribing for respiratory tract infections; respiratory tract infections
MeSH Terms: conditions — Pneumonia; Virus Diseases; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antimicrobial Stewardship Bundle (Experimental): An intervention "bundle" to reduce outpatient antibiotic use in children will include education, creation of and access to guidelines, and audit of and feedback on individual prescribing within the context of achievable benchmarks.
  Interventions: Behavioral: Antimicrobial Stewardship Bundle
- Control (No Intervention): Control sites will be within strata to maintain balance of treatment arm within strata

INTERVENTIONS:
Behavioral: Antimicrobial Stewardship Bundle — Guidelines, Education, Audit and Feedback
  Arms: Antimicrobial Stewardship Bundle

SUMMARY:
The purpose of the study is to determine if physician education coupled with audit and feedback of antibiotic prescribing can improve antibiotic prescribing by primary care clinicians.

DETAILED DESCRIPTION:
Using a large, diverse pediatric primary care network sharing a comprehensive electronic health record (EHR), a cluster-randomized trial will be performed to determine the effectiveness of an outpatient antimicrobial stewardship bundle, including treatment guidelines coupled with audit and feedback of physician prescribing, to curb inappropriate antibiotic prescribing for respiratory tract infections.

Aim 1: To determine the impact of an outpatient antimicrobial stewardship bundle within a pediatric primary care network on antibiotic prescribing for conditions for which antibiotics are not indicated.

Hypothesis: Antimicrobial stewardship will decrease rates of antibiotic prescribing for conditions for which antibiotics are not indicated.

Aim 2: To determine the impact of an outpatient antimicrobial stewardship bundle within a pediatric primary care network on broad-spectrum antibiotic prescribing for conditions for which narrow-spectrum antibiotics are indicated.

Hypothesis: Antimicrobial stewardship will decrease the rate of broad-spectrum antibiotic prescribing for conditions for which narrow-spectrum antibiotics are indicated.

ELIGIBILITY:
Inclusion Criteria:

* Primary care pediatric practices within the CHOP Care Network

Exclusion Criteria:

* Academic primary care pediatric practices within the CHOP Care Network
* Providers entering a practice after the start of the intervention
* Providers with less than 25 antibiotic prescriptions in the 6 months prior to the start of the intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reduction in the rate of broad-spectrum antibiotic prescribing for targeted conditions for which narrow-spectrum antibiotic therapy is indicated | from 20 months prior through 13 months post intervention
  The primary outcome measure seeks to determine if the incorporation of treatment guidelines coupled with audit and feedback of physician prescribing can reduce the the rate of antibiotic prescribing for targeted conditions for which antibiotic therapy is not indicated.

SECONDARY OUTCOMES:
The rate of antibiotic prescribing for targeted conditions for which antibiotic therapy is not indicated | from 20 months prior through 13 months post intervention
  The secondary outcome measure seeks to determine the rate of broad-spectrum antibiotic prescribing for targeted conditions for which narrow-spectrum antibiotic therapy is indicated. Thus, two classes of diagnoses will be collected: 1) respiratory tract infections for which no antibiotics are indicated, represented by a group codes indicating common infections with presumed viral etiology and 2) bacterial respiratory tract infections for which narrow spectrum antibiotics are indicated

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Gerber, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gerber JS, Prasad PA, Fiks AG, Localio AR, Bell LM, Keren R, Zaoutis TE. Durability of benefits of an outpatient antimicrobial stewardship intervention after discontinuation of audit and feedback. JAMA. 2014 Dec 17;312(23):2569-70. doi: 10.1001/jama.2014.14042. No abstract available. PMID 25317759
- [Derived] Gerber JS, Prasad PA, Fiks AG, Localio AR, Grundmeier RW, Bell LM, Wasserman RC, Keren R, Zaoutis TE. Effect of an outpatient antimicrobial stewardship intervention on broad-spectrum antibiotic prescribing by primary care pediatricians: a randomized trial. JAMA. 2013 Jun 12;309(22):2345-52. doi: 10.1001/jama.2013.6287. PMID 23757082